CLINICAL TRIAL: NCT04261192
Title: Establishment of Squamous Cell Organoids of the Head and Neck to Assess Their Response to Innovative Therapies
Acronym: ORGAVADS
Status: Recruiting | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A03332-55
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Organoid
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Constitution of tumor and blood samples — Constitution of tumor and blood samples

SUMMARY:
The emergence of tumor organoid cultures in recent years has made it possible to widen the repertoire of available preclinical tumor models and to bridge the gap between cell lines and tumors of xenografted patients in mice (PDXs).These organoids have the advantages of being able to be amplified fairly quickly after resection of the tumor, of having unlimited proliferation potential, a high rate of establishment success, and the possibility of being transfected and cryopreserved. These characteristics therefore allow them to summarize the clinical spectra of cancers, but also to be models for studying tumor progression as has been done with organoids for colorectal cancer. They are also very close morphologically and genetically to the tumor from which they derive.Finally, clinical trials are underway to determine whether the organoids of mammary, pulmonary and colorectal cancers can predict the response to patients' treatments and guide the therapeutic decision.It would therefore be possible to test multiple treatments on different samples. This would allow screening of a panel of treatments on a given tumor type but also to test a treatment ex vivo before administering it to the patient in vivo. This prospect is very interesting in particular in the tumors of the VADS where more than two thirds of the operated patients will benefit from a complementary treatment by radiotherapy and / or chemotherapy whose consequences can be important. Despite this adjuvant management, up to 30% of patients will relapse, highlighting a variable tumor chemosensitivity. This screening could make it possible to refine the choice of treatments adapted to each patient and thus limit the undesirable effects.The feasibility of establishing head and neck squamous cell organoid lines seems encouraging, with organoids derived from squamous cell carcinoma of the oral cavity and oropharynx having been recently established.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Patient with squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, classified T3Nx or T4Nx or T2N +, not previously treated;
* Patient to be treated by surgery;
* Patient affiliated to a social security scheme;
* No opposition to participate in the study

Exclusion Criteria:

* Pregnant woman ;
* Persons deprived of their liberty or under guardianship (including curatorship);
* History of malignant pathology preceding inclusion (apart from basal cell carcinomas of the skin and carcinomas in situ of the cervix treated surgically) or concomitant at inclusion (synchronous tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, classified T3Nx or T4Nx or T2N +, not previously treated;
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Rate of establishment of exploitable organoids tumor | 5 years
  Number of exploitable organoids tumor

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - CHU de Caen, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perreard M, Florent R, Divoux J, Grellard JM, Lequesne J, Briand M, Clarisse B, Rousseau N, Lebreton E, Dubois B, Harter V, Lasne-Cardon A, Drouet J, Johnson A, Le Page AL, Bazille C, Jeanne C, Figeac M, Goardon N, Vaur D, Micault E, Humbert M, Thariat J, Babin E, Poulain L, Weiswald LB, Bastit V. ORGAVADS: establishment of tumor organoids from head and neck squamous cell carcinoma to assess their response to innovative therapies. BMC Cancer. 2023 Mar 9;23(1):223. doi: 10.1186/s12885-023-10692-x. PMID 36894916